CLINICAL TRIAL: NCT01769274
Title: A RANDOMIZED, DOUBLE BLIND THIRD PARTY OPEN PLACEBO-CONTROLLED EXPLORATORY STUDY TO EVALUATE THE EFFICACY AND SAFETY OF SINGLE DOSES OF PF-05089771 IN PATIENTS WITH PRIMARY (INHERITED) ERYTHROMELALGIA
Brief Title: Evaluation Of The Efficacy And Safety Of Single Doses Of PF-05089771 In Patients With Primary (Inherited) Erythromelalgia
Acronym: IEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B3291006
Record Dates: First submitted 2012-10-18; First posted 2013-01-16 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Inherited Erythromelalgia
MeSH Terms: interventions — PF-05089771

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05089771 1600 mg (Experimental)
  Interventions: Drug: PF-05089771
- Placebo comparator: matching placebo (Placebo Comparator): Single oral dose of placebo for PF-05089771 1600 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05089771 — A single oral dose of PF-05089771 1600 mg solution to be administered on Day 1 of each treatment session. There are 2 treatment sessions, therefore 2 single oral doses of PF-05089771 will be adminstered.
  Arms: PF-05089771 1600 mg
Drug: Placebo — Placebo for PF-05089771 1600 mg solution administered in each treatment session. There are 2 treatment sessions, therefore 2 single oral doses of placebo will be administered.
  Arms: Placebo comparator: matching placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of single doses of PF-05089771 against placebo in treatment of pain in patients with primary, inherited erythromelalgia.

ELIGIBILITY:
Inclusion Criteria:

* Male and or female subjects between the ages of 18-78 years
* Subject has clinical signs of IEM
* Minimum BMI 17.5kg/m2 and total body weight >50kg

Exclusion Criteria:

* Other severe pain conditions, e.g. rheumatologic, that may impair subject's self-assessment of pain due to IEM.
* Evidence of clinically significant hypertension, clinically significant hematological, dermatological, renal, endocrine (except diabetes mellitus), pulmonary, gastrointestinal, cardiovascular, hepatic, neurological (other than IEM), or allergic disease (including drug allergies but excluding untreated asymptomatic seasonal allergies).
* Subjects with severe obesity.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10-22 (Actual); Primary Completion 2013-07-12 (Actual); Study Completion 2013-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cao L, McDonnell A, Nitzsche A, Alexandrou A, Saintot PP, Loucif AJ, Brown AR, Young G, Mis M, Randall A, Waxman SG, Stanley P, Kirby S, Tarabar S, Gutteridge A, Butt R, McKernan RM, Whiting P, Ali Z, Bilsland J, Stevens EB. Pharmacological reversal of a pain phenotype in iPSC-derived sensory neurons and patients with inherited erythromelalgia. Sci Transl Med. 2016 Apr 20;8(335):335ra56. doi: 10.1126/scitranslmed.aad7653. PMID 27099175
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291006&StudyName=%20Evaluation%20Of%20The%20Efficacy%20And%20Safety%20Of%20Single%20Doses%20Of%20PF-05089771%20In%20Patients%20With%20Primary%20%28Inherited%29%20Erythromelalgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Participants were exposed to pain stimulus. Reproducibility and repeatability of induced pain attacks and spontaneous reporting of pain by participants was established. Part A was performed for 1-2 days and maximum up to 7 days. Maximum duration between Part A and Part B was of 4 weeks.
- Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771: On completion of Part A, participants were randomized in Part B. Part B: Participants were randomized to receive oral dispersion of PF-05089771 1600 milligram (mg) on Day 1 of Treatment session 1 (Study Period 1), followed by washout of 72 hours. Then, participants received oral dispersion of placebo matched to PF-05089771 on Day 5 of Treatment session 1 (Study Period 2). Treatment session 1 was followed by washout of 72 hours and then Treatment session 2. On Day 1 of Treatment session 2 (Study Period 3), participants received oral dispersion of placebo matched to PF-05089771, followed by washout of 72 hours. Then, participants received oral dispersion of PF-05089771 1600 mg on Day 5 of Treatment session 2 (Study Period 4). Maximum permitted interval between Study Period 2 completion and the start of Study Period 3 is 6 months.
- Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo: On completion of Part A, participants were randomized in Part B. Part B: Participants were randomized to receive oral dispersion of placebo matched to PF-05089771 on Day 1 of Treatment session 1 (Study Period 1), followed by washout of 72 hours. Then, participants received oral dispersion of PF-05089771 1600 mg on Day 5 of Treatment session 1 (Study Period 2). Treatment session 1 was followed by washout of 72 hours and then Treatment session 2. On Day 1 of Treatment session 2 (Study Period 3), participants received oral dispersion of PF-05089771 1600 mg, followed by washout of 72 hours. Then, participants received oral dispersion of placebo matched to PF-05089771 on Day 5 of Treatment session 2 (Study Period 4). Maximum permitted interval between Study Period 2 completion and the start of Study Period 3 is 6 months.
Period: Part A
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B:Treatment Session1-Period1
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Part B:Treatment Session1-Period2
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Part B:Treatment Session2-Period3
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Part B:Treatment Session2-Period4
Arm/Group | Part A | Part B: PF-05089771 Then Placebo Then Placebo Then PF-05089771 | Part B: Placebo Then PF-05089771 Then PF-05089771 Then Placebo
Started | 0 | 2 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of study medication.
Groups:
- All Participants: All participants who were enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity Numerical Rating Scale (PI-NRS) Score - From 0 to 4 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10, where 0= no pain and 10= worst possible pain; higher scores signify more pain. The average pain score was calculated as the mean of the pain scores recorded every 15 minutes from 0 to 4 hours post-dose.
Time Frame: Every 15 minutes from 0 to 4 hours post-dose
Population: Full analysis set included all participants who successfully completed Part A, were randomized in Part B, and who received at least 1 dose of randomized study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Treatment Session 1: PF-05089771 1600 mg: Participants received oral dispersion of PF-05089771 1600 mg in Treatment session 1.
- Treatment Session 1: Placebo: Participants received oral dispersion of placebo matched to PF-05089771 in Treatment session 1.
- Treatment Session 2: PF-05089771 1600 mg: Participants received oral dispersion of PF-05089771 1600 mg in Treatment session 2.
- Treatment Session 2: Placebo: Participants received oral dispersion of placebo matched to PF-05089771 in Treatment session 2.
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Units on a scale | 2.08 (2.20) | 2.73 (2.68) | 1.95 (2.29) | 2.04 (1.81)

2. Secondary Outcome: Average PI-NRS Score - From Post Evoked Pain Time Point 2 (EP2) to 8 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 2= first time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP2 is approximately a time point 4-5 hours post-dose. The average pain score was calculated as the mean of the pain scores recorded from EP2 to 8 hours post-dose.
Time Frame: Post EP2, every 5 minutes for the first hour, then every 15 minutes up to 8 hours post-dose
Population: Full analysis set included all participants who successfully completed Part A, were randomized in Part B, and who received at least 1 dose of randomized study medication. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
Units on a scale | 0.70 (0.64) | 0.61 (0.46) | 0.55 (0.51) | 1.08 (0.63)

3. Secondary Outcome: Average PI-NRS Scores - From Post Evoked Pain Time Point 3 (EP3) to 10 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 3= second time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP3 is approximately a time point 8-9 hours post-dose. The average pain score was calculated as the mean of the pain scores recorded from EP3 to 10 hours post-dose.
Time Frame: Post EP3, every 5 minutes for the first hour, then every 15 minutes up to 10 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
Units on a scale | 1.19 (1.22) | 1.55 (1.15) | 0.82 (0.52) | 1.39 (0.58)

4. Secondary Outcome: Average PI-NRS Scores - From Post Evoked Pain Time Point 4 (EP4) to 28 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 4= third time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP4 is approximately a time point 24-25 hours post-dose. The average pain score was calculated as the mean of the pain scores recorded from EP4 to 28 hours post-dose.
Time Frame: Post EP4, every 5 minutes for the first hour, then every 15 minutes up to 28 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3
Units on a scale | 0.99 (0.52) | 0.91 (0.53) | 0.36 (0.08) | 0.77 (0.38)

5. Secondary Outcome: Maximum PI-NRS Scores - From 0 Hour to 4 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Maximum pain score in 4 hours period post-dosing is reported.
Time Frame: From 0 hour to 4 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Units on a scale | 7.6 (1.7) | 8.0 (1.4) | 8.2 (2.1) | 8.6 (1.1)

6. Secondary Outcome: Maximum PI-NRS Scores - From Post EP2 to 8 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 2= first time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP2 is approximately a time point 4-5 hours post-dose. Maximum pain score in period from post EP2 to 8 hours post-dose is reported.
Time Frame: From post EP2 to 8 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
Units on a scale | 3.5 (1.7) | 5.7 (3.1) | 5.5 (3.3) | 7.8 (1.9)

7. Secondary Outcome: Maximum PI-NRS Scores - From Post EP3 to 10 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 3= second time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP3 is approximately a time point 8-9 hours post-dose. Maximum pain score in period from post EP3 to 10 hours post-dose is reported.
Time Frame: From the end of EP3 to 10 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
Units on a scale | 2.3 (2.6) | 6.0 (3.6) | 5.3 (2.6) | 8.3 (2.1)

8. Secondary Outcome: Maximum PI-NRS Scores - From Post EP4 to 28 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 4= third time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP4 is approximately a time point 24-25 hours post-dose. Maximum pain score in period from post EP4 to 28 hours post-dose is reported.
Time Frame: Post EP4, every 5 minutes for the first hour, then every 15 minutes up to 28 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3
Units on a scale | 7.3 (1.2) | 7.3 (2.5) | 5.7 (2.1) | 8.0 (2.0)

9. Secondary Outcome: Duration When PI-NRS Scores Were Greater Than (>) 5 - From 0 Hour to 4 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. The duration of time that participants experienced PI-NRS score greater than 5 from the 0 hours to 4 hours post-dose.
Time Frame: From 0 hour to 4 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Minutes | 20.0 (42.0) | 29.4 (63.0) | 10.4 (23.3) | 8.2 (12.1)

10. Secondary Outcome: Duration When PI-NRS Scores Were >5 - From Post EP2 to 8 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 2= first time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP2 is approximately a time point 4-5 hours post-dose. The duration of time that participants experienced PI-NRS score >5 from in period from post EP2 to 8 hours post-dose is reported.
Time Frame: Post EP2, every 5 minutes for the first hour, then every 15 minutes up to 8 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
Minutes | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

11. Secondary Outcome: Duration When PI-NRS Scores Were >5 - From Post EP3 to 10 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 3= second time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP3 is approximately a time point 8-9 hours post-dose. The duration of time that participants experienced PI-NRS score >5 from the post EP3 to 10 hours post dose.
Time Frame: Post EP3, every 5 minutes for the first hour, then every 15 minutes up to 10 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
Minutes | 0.0 (0.0) | 0.0 (10.4) | 0.0 (0.0) | 0.0 (0.0)

12. Secondary Outcome: Duration When PI-NRS Scores Were >5 - From Post EP4 to 28 Hours Post-dose
Description: Participants rated severity of their pain at 11 point PI-NRS, by choosing a number between 0 and 10. Where 0= no pain and 10= worst possible pain; higher scores signify more pain. Evoked pain time point 4= third time point post-dose when pain was evoked using the participant specific heat pain stimulus. EP4 is approximately a time point 24-25 hours post-dose. The duration of time that participants experienced PI-NRS score >5 from post EP4 to 28 hours post-dose.
Time Frame: After EP4, every 5 minutes for the first hour, then every 15 minutes up to 28 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3
Minutes | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

13. Secondary Outcome: Number of Participants With Participant's Global Satisfaction Score
Description: Participant was asked "How would you rate the study medication you received for pain?". The participant was provided the following choices as an answer: excellent=4; good=3; fair=2; poor=1. Response to this question, was participant's overall impression (global evaluation) of the study medication at 4 hour post-dose or at time of first rescue treatment or medication, which ever occurred first.
Time Frame: At 4 hour post-dose or at time of first rescue therapy, whichever occurred first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants
  Poor Score | 1 | 3 | 0 | 4
  Fair Score | 2 | 1 | 3 | 1
  Good Score | 1 | 0 | 1 | 0
  Excellent Score | 1 | 1 | 1 | 0

14. Secondary Outcome: Time to First Use of Rescue Therapy or Medication
Description: Time to rescue medication (hour) was calculated as: date/time of rescue medication minus date/time of first dose for each period. If participant who did not receive rescue medication, the time of censoring was cut off at 24 hours or the time of withdrawal, whichever was earlier. Kaplan-Meier method was used for estimation.
Time Frame: Up to maximum of 24 hours post-dose
Population: Full analysis set included all participants who successfully completed Part A, were randomized in Part B, and who received at least 1 dose of randomized study medication. Number of Participants Analyzed = number of participants evaluable for this outcome measure.
Measure: Mean (90% Confidence Interval); unit: Hours
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 2
Hours | 14.9 [1.6 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants. | 2.3 [1.8 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants. | 15.3 [1.6 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants. | 10.3 [1.5 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants.
Statistical Analysis 1: Comparison: Treatment Session 1: PF-05089771 1600 mg vs Treatment Session 1: Placebo; Test type: Other; p = 1.0000, Hierarchical rank test
Statistical Analysis 2: Comparison: Treatment Session 2: PF-05089771 1600 mg vs Treatment Session 2: Placebo; Test type: Other; p = 1.0000, Hierarchical rank test

15. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the 24 Hour Post-dose (AUC24) of PF-05089771
Time Frame: Predose, 0.5, 2, 4, 6, and 24 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis set included all participants who were randomized, received study medication, and had at least 1 of the PK parameters of interest in at least 1 treatment session.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 2: PF-05089771 1600 mg
Number analyzed (Participants) | 5 | 5
Nanogram*hour per milliliter (ng*hr/mL) | 652100 (19) | 657500 (26)

16. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-05089771
Time Frame: Predose and 0.5, 2, 4, 6, and 24 hours post dose
Population: PK parameter analysis set included all participants who were randomized, received study medication, and had at least 1 of the PK parameters of interest in at least 1 treatment session.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 2: PF-05089771 1600 mg
Number analyzed (Participants) | 5 | 5
Nanogram*hour per milliliter (ng*hr/mL) | 652400 (19) | 658000 (26)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05089771
Time Frame: Predose and 0.5, 2, 4, 6, and 24 hours post dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 2: PF-05089771 1600 mg
Number analyzed (Participants) | 5 | 5
Nanogram per milliliter (ng/mL) | 66760 (22) | 59080 (21)

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05089771
Time Frame: Predose and 0.5, 2, 4, 6, and 24 hours post dose
Population: as for outcome 16
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 2: PF-05089771 1600 mg
Number analyzed (Participants) | 5 | 5
Hours | 3.95 [2.00 to 6.07] | 6.00 [4.00 to 6.13]

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state.
Time Frame: Baseline up to a maximum of Day 83
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants
  AEs | 5 | 5 | 5 | 4
  SAEs | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory abnormalities: Hemoglobin (Hgb), hematocrit, red blood cell count: less than(<)0.8*lower limit of normal(LLN), platelet: <0.5*LLN/greater than (>)1.75*upper limit of normal (ULN), white blood cell: <0.6*LLN/>1.5*ULN, lymphocyte, neutrophil (absolute, %):<0.8*LLN/>1.2*ULN, total neutrophil <0.8*LLN;basophil, eosinophil, monocyte (absolute, %):>1.2*ULN; mean corpuscular (MC) volume, mean cell hemoglobin, MC hemoglobin concentration, mean platelet volume: <0.9*LLN/>1.1*ULN; total bilirubin >1.5*ULN, aspartate aminotransferase (AT), alanine AT, gammaglutamyl transferase, alkaline phosphatase:> 3.0*ULN, total protein, albumin: <0.8*LLN/>1.2*ULN; blood urea nitrogen, creatinine:>1.3*ULN, uric acid >1.2*ULN; sodium <0.95*LLN/>1.05*ULN, potassium, chloride, calcium, magnesium, bicarbonate: <0.9*LLN/>1.1*ULN; glucose <0.6*LLN/>1.5*ULN; urine (specific gravity <1.003/>1.030, pH <4.5/>8, glucose, ketone, protein, blood/Hgb, urobilinogen, bilirubin, nitrite, leukocyte esterase >=1).
Time Frame: Baseline up to a maximum of Day 73
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 2 | 2 | 2 | 2

21. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Core Body Temperature
Description: The minimum starting temperature to measure core body temperature used was 33 degree Celsius. Clinically significant changes from baseline in core body temperature was judged by investigator.
Time Frame: Baseline up to a maximum of Day 83
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Blood Pressure
Description: Criteria for clinically significant blood pressure abnormalities: systolic blood pressure >=30 millimetre of Mercury (mmHg) change from baseline in same posture, systolic blood pressure <90 mmHg, diastolic blood pressure >=20 mmHg change from baseline in same posture, diastolic blood pressure <50 mmHg.
Time Frame: Baseline up to a maximum of Day 83
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Electrocardiogram (ECG)
Description: Criteria for clinically significant abnormalities in ECG : PR interval >=300 millisecond (msec) and 25 percent (%) increase when baseline >200 msec, 50% increase when baseline less than or equal to (<=) 200 msec; QRS interval >=140 msec, >=50% increase from baseline; QT interval >=500 msec; QT interval corrected using the Fridericia formula (QTcF) 450 msec to <480 msec, >=480 msec, 30 to <60 msec increase from baseline, >=60 msec increase from baseline.
Time Frame: Baseline up to a maximum of Day 83
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study. Adverse events were collected only for Part B of the study.
Arm/Group | Treatment Session 1: PF-05089771 1600 mg | Treatment Session 1: Placebo | Treatment Session 2: PF-05089771 1600 mg | Treatment Session 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Session 1: PF-05089771 1600 mg (N=5) | Treatment Session 1: Placebo (N=5) | Treatment Session 2: PF-05089771 1600 mg (N=5) | Treatment Session 2: Placebo (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 4 | 0 | 3 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 1
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 3 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 4 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.